CLINICAL TRIAL: NCT01624688
Title: Optimizing Tattoo Removal: a Side-by-side Comparison in the Search for One Treatment Tattoo Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Professor Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011P001091
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Tattoo; Tattoo Removal
Keywords: Tattoo; Tattoo Removal
MeSH Terms: interventions — Tattoo Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Tattoo Removal — Tattoo removal with q-switched laser treatment, repeated q-switched laser treatment, repeated q-switched laser treatment with fractional ablative laser treatment, and repeated q-switched laser treatment with fractional ablative laser treatment and then topical urea

SUMMARY:
The purpose of this study is to combine treatment options for tattoo removal in an attempt to completely remove a tattoo in one visit.

DETAILED DESCRIPTION:
Efficient tattoo removal is of special concern to dermatology, where tattoo removal is a common request. Current tattoo removal techniques using once monthly treatment with quality-switched (QS) lasers are relatively effective, but not efficient. Numerous treatments are required and complete removal of ink is usually rare, making the process time-consuming, expensive and, sometimes, disappointing. The broad objective of this study is to combine effective methods for tattoo removal based on current knowledge to establish a protocol which significantly improves laser tattoo removal, aiming to selectively remove most tattoos in one office visit.

The proposed study is a prospective, side-by-side comparison of four tattoo treatment protocols using a combination of ablative fractional and q-switched (QS) laser techniques. 32 subjects with tattoos recruited from the community will receive all four treatments, one on each randomly-assigned, equal quadrant of the same tattoo. The different treatment protocols are as follows: 1. one round of QS laser treatment, which is the current treatment standard 2. four repeat treatments with the QS laser with a 20 minute delay in between 3. four repeat treatments at 20 minute intervals with the QS laser combined with an ablative fractional laser treatment 4. four repeat treatments at 20 minute intervals with the QS laser plus treatment with the ablative fractional laser, in combination with topical urea application. Following this initial round of treatments, the subject will have the option to choose his or her preferred treatment protocol which will then be used to treat the entire tattoo again one month later. Previous studies indicate that the majority of tattoos will be completely or nearly completely removed in this study, providing a potential benefit to those who enroll in the study. The primary measures of efficacy are (a) blinded evaluation of improvement from standard digital photographs taken before and after the treatments, including number of tattoos that are completely gone, and (b) digital analysis of tattoo removal from those photos. Other study endpoints include patient's preferred removal technique, evaluation of tattoo ink on dressings, inflammatory and pigmentary alterations and changes in skin texture.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 18 and 50 years old, male or female.
* Subjects with tattoos that are between 16 and 400 cm2, both amateur and professional
* Willingness to participate in the study
* Willingness to shield tattoo completely from sun exposure
* Willingness to receive EXPERIMENTAL treatment
* Informed consent agreement signed by the subject
* Willingness to follow the treatment schedule and post treatment care requirements

Exclusion Criteria:

* Subjects with recent sun exposure and suntan in the area to be treated
* Allergic tattoos (hypersensitivity to tattoo ink)
* History of vitiligo
* Tattoos located on the neck or face
* Subjects unwilling to tolerate partial removal of the tattoo in this study
* Infection or skin disease in the area to be treated
* Subjects who are immunosuppressed
* Subject is unable to comply with treatment, home care or follow-up visits
* Subject is pregnant or nursing
* Allergy to lidocaine
* Liver failure

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Tattoo Clearance | 2 months after treatment

SECONDARY OUTCOMES:
Patient's preferred removal technique | 2 months after treatment
Post treatment skin changes | 2 months after treatment
  inflammatory and pigmentary alterations and changes in skin texture after treatment

CONTACTS AND LOCATIONS:
Overall Officials: R. Rox Anderson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Wellman Center for Photomedicine, Boston, Massachusetts, United States